CLINICAL TRIAL: NCT05035290
Title: Negative Pressure Ventilation in Critically Ill Paediatric Patients During Weaning: Prospective Randomized Interventional Trial
Brief Title: Negative Pressure Ventilation in Paediatric Patients During Weaning
Acronym: NEGWEAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KDAR NEGATIVE
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Weaning Failure
Keywords: Weaning; Weaning failure; Negative pressure ventilation; Cuirass; Paediatric patient; Critical care

STUDY DESIGN:
Intervention Model Description: Critically ill paediatric patients scheduled for weaning from mechanical ventilation will be randomized to interventional group (negative pressure ventilation) and control group (standard approach)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative pressure ventilation (Experimental): Negative pressure application after extubation
  Interventions: Device: Negative pressure ventilation
- Standard approach (No Intervention): Standard approach - oxygentherapy based on patients need

INTERVENTIONS:
Device: Negative pressure ventilation — Negative pressure ventilation - cuirass will be applied on the patient´s ches and abdomen immediately after extubation
  Other Names: Negative pressure ventilation - cuirass
  Arms: Negative pressure ventilation

SUMMARY:
Negative pressure ventilation (NPV) represent a unique form of noninvasive ventilation using negative pressure by specialized cuirass, that evolve negative pressure on the front size of chest and partially abdomen and facilitate the spontaneous breathing. The benefit of NPV beside noninvasive application, is the supreme tolerance of the patient (compared to other forms of noninvasive ventilation - mask, helmet), without the negative impact on enteral feeding tolerance and with the possibility of active physiotherapy. NPV could be even combined with oxygentherapy or noninvasive positive pressure ventilation. NPV in paediatric patients after extubation could be associated with reduced incidence of weaning failure.

DETAILED DESCRIPTION:
After ethics committee approval and informed consent from legal guardians and fulfilling inclusion criteria, critically ill paediatric patients scheduled for weaning will be randomized (in 1:1 allocation) to NPV (interventional group) or standard approach (without NPV) after extubation. NPV in paediatric patients after extubation could be associated with reduced incidence of weaning failure. The initial setting on NPV will be: negative pressure set to -10cmH2O and will proceed for minimal time of 60 minutes after extubation (will proceed longer in case of good tolerance). In case of hypoxaemia, additional oxygentherapy will be administered according to the patients condition Primary outcome will be defined as postextubation failure incidence at 60 minutes after extubation (defined as need of noninvasive positive pressure ventilation, intubation, or high-flow oxygen therapy) and the overall incidence of weaning failure during initial 24 hour after extubation. The secondary outcome will be the dynamics of blood gases (arterial or capillary blood sample) during initial 60 minutes after extubation (1. extubation, 2. 60 minutes after extubation) and the need of and amount of artificial oxygentherapy (litres of oxygen per minute, pulse oximetry). Another outcome will be the overall cuirass tolerance after 60 minutes and after 24 hours defined by incidence of skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* invasive mechanical ventilation
* informed consent
* scheduled for weaning

Exclusion Criteria:

* neuromuscular disorder
* mechanical ventilation at home (chronic use)
* less than 24 hours after abdominal or thoracic surgery
* technical problems with the cuirass - chest drain

Ages: 1 Month to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Early weaning failure | in 60 minutes after extubation
  Incidence of early weaning failure - intubation, noninvasive positive pressure ventilation, high flow oxygen therapy
Overall weaning failure | during 24 hours after extubation
  Incidence of weaning failure - intubation, noninvasive positive pressure ventilation, high flow oxygen therapy

SECONDARY OUTCOMES:
Blood gases trends | during initial 60 minutes after extubation
  Trends of blood gases (CO2 and O2) in arterial or capillary blood samples drown at the extubation and in 60 minutes after extubation
Pulse oximetry trend | during initial 60 minutes after extubation
  Trends of pulse oximetry during initial 60 minutes after extubation
Early cuirass tolerance | during initial 60 minutes after extubation
  Incidence of the need for cuirass removal during initial 60 minutes
Overall cuirass tolerance | during 24 hours after extubation
  Defined by incidence of new skin lesions after cuirass application

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided